CLINICAL TRIAL: NCT07001969
Title: Massoud-Goel Technique and Theory: Percutaneous Trans-facet Fixation for Treatment of Degenerative Spine
Brief Title: Percutaneous Trans-facet Spine Fixation
Acronym: Massoud-Goel
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Massoud (Other)
Collaborators: Cairo University (Other); Military Academy for Medical Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Mahmoud Massoud, Lecturer Orthopedic surgery department Orthopedic Surgery AFCM Cairo Egypt, Consultant spine surgery Helmya Military hospital, Spine unit., Armed Forces College of Medicine, Cairo, Egypt
Organization: Armed Forces College of Medicine, Cairo, Egypt (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGY-2025-PTFF-MGT-001
Record Dates: First submitted 2025-02-13; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Spine; Degeneration of Lumbar Intervertebral Disc; Degenerative Cervical Disc Disease; Ligamentum Flavum Hypertrophy; Spinal Canal Stenosis; Spine Instability
Keywords: Percutaneous; Trans-facet; Fixation; Massoud-Goel; Technique and Theory for Treatment of Degenerative Spine
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Percutaneous Trans-Facet Fixation Using the Massoud-Goel Technique and Theory for Degenerative Spine (Experimental): This study arm involves the use of Percutaneous Trans-Facet Fixation (PTFF) with the Massoud-Goel Technique and Theory (MGT) for the treatment of degenerative spine conditions, Looking for signs of instability. In this arm will undergo minimally invasive trans-facet screw fixation to provide spinal stability while preserving mobility and reducing soft tissue disruption.
  The intervention includes:
  * Preoperative Assessment: MRI and CT scans to evaluate facet joint degeneration and spinal instability.
  * Surgical Technique: Percutaneous placement of facet screws under fluoroscopic guidance, following the principles of the Massoud-Goel Technique.
  * Postoperative Care: Patients will follow a structured rehabilitation program, including pain management and physiotherapy, to assess functional recovery and long-term outcomes.
  The study aims to evaluate radiological fusion rates, pain relief (VAS scores), functional improvement (ODI scores), and complication rates associations.
  Interventions: Procedure: Massoud-Goel Technique and Theory; Procedure: Percutaneous Trans-facet Fixation for Treatment of Degenerative Spine

INTERVENTIONS:
Procedure: Massoud-Goel Technique and Theory — Percutaneous Trans-facet Fixation Massoud-Goel Technique and Theory for Treatment of Degenerative Spine
Procedure: Percutaneous Trans-facet Fixation for Treatment of Degenerative Spine — Percutaneous Trans-facet Fixation (Developmental of Dr Atul goel technique of transfacet fixation by open surgery using Magrel technique) Massoud-Goel Technique and Theory for Treatment of Degenerative Spine

SUMMARY:
Percutaneous Trans-facet Fixation Massoud-Goel Technique and Theory for Treatment of Degenerative Spine

DETAILED DESCRIPTION:
Massoud-Goel' as rationale treatment for treatment spinal degeneration affected spinal segments using trans-articular screws, without physically distracting the facets, or removal of any part of the bone or ligament.

Following fixing of the segment, all the secondary phenomenon reverse, effectively increasing the canal size and reversing the effects of spinal degeneration and spinal canal stenosis.

Stabilizes the region and provides an environment for resorption of the herniated disc and ultimate arthrodesis of the spinal segments.

ELIGIBILITY:
Inclusion Criteria:

For Lumbar Sub-axial cervical instability Clinical radicular symptoms can indicate the level of spinal instability. The presence of osteophytes. Reduction of the intervertebral disc space. Disc prolapse. Ligamentum flavum buckling. For atlantoaxial instability Cervical myelopathy clinical Alteration of atlantodental interval on dynamic flexion-extension images.

Exclusion Criteria:

1. Cauda equine syndrome
2. Progressive motor weakness
3. Failed damage control method
4. Spondylolisthesis, Spondyolysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 3 months
  Relief of pain from neuralgia (sciatica & brachialgia) also claudication pain assessment by visual analogue scale 1-10

SECONDARY OUTCOMES:
Functional recovery | 3 months
  functional improvement postoperatively. Secondary outcomes include functional recovery (Oswestry Disability Index score)
Less complications | 1 year
  fusion rates (CT scan), and complication rates, assessing both efficacy and safety.
  Additional measures like hospital stay duration and patient satisfaction provide insights into procedural efficiency and patient-reported outcomes.
Spinal stability | 6 months
  By CT spine we can assess facet fusion, stabilization of spine segmental instability
Neurological decompression indirectly | 6 months
  Early by position of patients intraoperative and stabilization, late by healing of pathological state of ligament flavum hypertrophic changes, disc degeneration, spinal canal stenosis by Magnetic resonance imaging follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- 434, Cairo, Shorouk, Egypt

IPD SHARING:
Plan to Share IPD: Yes
New researches
Supporting Information: Study Protocol
Time Frame: 7 years
Access Criteria: IPD Sharing Access Criteria for the Study:**
  **"Percutaneous Trans-Facet Fixation Using the Massoud-Goel Technique for Treatment of Degenerative Spine"
  1. Data Availability:
     * De-identified Individual Participant Data (IPD) will be made available for academic and research purposes.
     * Shared data will include patient demographics, radiographic outcomes, clinical assessments (VAS, ODI scores), and surgical parameters**.
  2. Access Requirements:
     * Researchers must submit a formal request with a brief research proposal outlining the intended use of the data.
     * Approval from an **Institutional Review Board (IRB) or Ethics Committee is mandatory.
     * A Data Use Agreement (DUA) must be signed to ensure compliance with ethical and legal regulations.
  3. Timing of Data Sharing:
     * Data will be available 6 months after the primary publication of study results.
     * The sharing period will extend for 5 years post-publ

REFERENCES:
- [Background] Borm W, Konig RW, Albrecht A, Richter HP, Kast E. Percutaneous transarticular atlantoaxial screw fixation using a cannulated screw system and image guidance. Minim Invasive Neurosurg. 2004 Apr;47(2):111-4. doi: 10.1055/s-2004-818449. PMID 15257485
- [Background] Magerl FP. Stabilization of the lower thoracic and lumbar spine with external skeletal fixation. Clin Orthop Relat Res. 1984 Oct;(189):125-41. PMID 6478690
- [Background] BOUCHER HH. A method of spinal fusion. J Bone Joint Surg Br. 1959 May;41-B(2):248-59. doi: 10.1302/0301-620X.41B2.248. No abstract available. PMID 13641310
- [Background] KING D. Internal fixation for lumbosacral fusion. J Bone Joint Surg Am. 1948 Jul;30A(3):560-5. No abstract available. PMID 18109577
- [Background] Goel A. Goel's classification of atlantoaxial "facetal" dislocation. J Craniovertebr Junction Spine. 2014 Jan;5(1):3-8. doi: 10.4103/0974-8237.135206. No abstract available. PMID 25013340
- [Background] Satoskar SR, Goel AA, Mehta PH, Goel A. Quantitative morphometric analysis of the lumbar vertebral facets and evaluation of feasibility of lumbar spinal nerve root and spinal canal decompression using the Goel intraarticular facetal spacer distraction technique: A lumbar/cervical facet comparison. J Craniovertebr Junction Spine. 2014 Oct;5(4):157-62. doi: 10.4103/0974-8237.147079. PMID 25558146
- [Background] Goel A. From "only decompression" to "only fixation:" A century-long journey of surgical treatment for spinal spondylosis. J Craniovertebr Junction Spine. 2018 Oct-Dec;9(4):219-220. doi: 10.4103/jcvjs.JCVJS_118_18. No abstract available. PMID 30783342
- See also: Collection of auther about the theory and the technique — https://t.me/drmassoud77/24301
- Available data/document: Individual Participant Data Set — https://t.me/drmassoud77/24301 — Book of author about technique